CLINICAL TRIAL: NCT05020275
Title: Relationship Between Resistance to the Tyrosine Kinase Inhibitor Osimertinib and Pharmacokinetics in Non-small Cell Lung Cancer: Toward an Individualization of the Treatment (RESISTYR)
Brief Title: Resistance to the Tyrosine Kinase Inhibitor Osimertinib and Pharmacokinetics in Non-small Cell Lung Cancer
Acronym: RESISTYR
Status: Active, not recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8892_RESISTYR
Record Dates: First submitted 2021-07-13; First posted 2021-08-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Non-small Cell Lung cancer; Osimertinib; Resistance; Pharmacokinetics
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Evaluate the influence of genetic polymorphisms on the plasma concentration of osimertinib (CYP3A4 and ABCB1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood samples: Blood samples for further assays
  Interventions: Diagnostic Test: Blood Samples

INTERVENTIONS:
Diagnostic Test: Blood Samples — * Samples for ctDNA blood concentration and osimertinib plasma concentration
  * Sample for genetic polymorphisms

SUMMARY:
Osimertinib is a tyrosine kinase (TKI) inhibitor targeting EGF-R (epidermal growth factor receptor) and used in the management of patients with non-small cell lung cancer (NSCLC) with oncogenic drug addiction to EGF-R. The results of the FLAURA study justifies this 3rd generation TKI as the first line TKI of choice since an increase in overall survival of several months has been observed compared to TKIs of previous generations (erlotinib, gefitinib). However, the response to osimertinib is heterogeneous and some patients are poor responder. In addition, even when an initial response to ITK is observed, the natural history of the disease inevitably leads to the appearance of resistance mutations and loss of efficacy of osimertinib after a few months of treatment.In the hypothesis of a concentration-effect relationship, an underexposure (an insufficient plasma concentration) to osimertinib could lead to a suboptimal response by favoring the appearance of molecular resistance. By analogy with the mechanisms of resistance to anti-infectives, the systemic concentration of TKI may have to be maintained above a certain value throughout the treatment to reach an effective concentration in the tumor, in order to to prevent the selection of resistant clones. The value of this approach for optimizing treatment with TKI has been shown for this therapeutic class. This mechanistic hypothesis has been suggested several TKIs.

In addition, the association between pharmacokinetics of TKIs and the development of resistance has been reported in several pilot studies for dasatinib, erlotinib. Furthermore, a link between TKI concentration and ctDNA concentration was demonstrated in a pilot study by Garlan et al. in 11 patients treated for melanoma with vemurafenib.

The impact of the results of this study is important since the aims are to identify preemptive and predictive biomarkers of drug response and to increase mechanistic knowledge regarding risk factor of resistance to osimertinib. Finally, if the hypotheses evaluated in this translational research study are verified, therapeutic drug monitoring of TKI (and ctDNA analysis) would be immediately applicable in clinical practice since the technical tools are already available in the laboratories of most hospitals centers.

DETAILED DESCRIPTION:
Osimertinib is a tyrosine kinase (TKI) inhibitor targeting EGF-R (epidermal growth factor receptor) and used in the management of patients with non-small cell lung cancer (NSCLC) with oncogenic drug addiction to EGF-R. The results of the FLAURA study justifies this 3rd generation TKI as the first line TKI of choice since an increase in overall survival of several months has been observed compared to TKIs of previous generations (erlotinib, gefitinib). However, the response to osimertinib is heterogeneous and some patients are poor responder. In addition, even when an initial response to ITK is observed, the natural history of the disease inevitably leads to the appearance of resistance mutations and loss of efficacy of osimertinib after a few months of treatment.

The occurrence of resistances is a major problem since they lead to treatment failure. Identifying biomarkers predictive of the response and / or the emergence of these mutations of resistance is therefore a research challenge. Indeed, knowing risk factors molecular resistance could help to optimize the treatment.

A first approach to monitor the disease is the measurment of residual disease circulating tumor DNA in the blood of patients (ctDNA). These minimally invasive "liquid biopsies" can be performed iteratively, unlike tissue biopsies. It is a dynamic biomarker with several advantages. On the one hand, it would be a biomarker for monitoring residual disease during treatment. The ctDNA concentration and its kinetics under treatment have also been associated with the clinical outcome. Better overall survival has thus been observed with the first generation molecules in patients with low baseline ctDNA concentration or a rapid decrease in the ctDNA concentration at the start of treatment. On the other hand, the analysis of ctDNA makes it possible to characterize the nature of the acquired resistance mutations appearing during treatment.

In addition, TKI are good candidates for therapeutic drug monitoring (TDM). The objective of TDM is to assess exposure by measuring plasma concentration. TKIs are characterized by interindividual pharmacokinetic (PK) variability. Indeed, taking into account their route of administration (per os) and their metabolism (substrate for CYP450 enzymes), plasma exposure is variable from one patient to another. Thus, at the same dosage, depending on absorption and metabolic capacity, patients are not likely to be exposed to the same plasma concentrations. This PK variability is also observed for osimertinib since interindividual coefficients of variation of plasma exposure of 50 to 60% have been reported.

In the hypothesis of a concentration-effect relationship, an underexposure (an insufficient plasma concentration) to osimertinib could lead to a suboptimal response by favoring the appearance of molecular resistance. By analogy with the mechanisms of resistance to anti-infectives, the systemic concentration of TKI may have to be maintained above a certain value throughout the treatment to reach an effective concentration in the tumor, in order to to prevent the selection of resistant clones. The value of this approach for optimizing treatment with TKI has been shown for this therapeutic class. This mechanistic hypothesis has been suggested several TKIs.

In addition, the association between pharmacokinetics of TKIs and the development of resistance has been reported in several pilot studies for dasatinib, erlotinib.

Furthermore, a link between TKI concentration and ctDNA concentration was demonstrated in a pilot study by Garlan et al. in 11 patients treated for melanoma with vemurafenib.

In NSCLC, it therefore appears relevant and innovative to study the relationship between the plasma concentration of osimertinib and the efficacy of the treatment. In addition, it would be relevant to investigate the correlation between the plasma concentration of osimertinib and ctDNA in order to assess whether osimertinib plasma exposure could be a risk factor of emergence of resistance to anti-EGF treatment. These two minimally invasive biomarkers could be integrated into a dynamic monitoring of the treatment response in a personalized medicine approach.

Results expected, perspectives As this is an observational study, there is no need to add invasive procedure compared to the usual follow-up of patients with NSCLC , the benefit / risk balance is favorable for the participants.

The expected benefit is collective since if the interest of a therapeutic follow-up by pharmacological (and oncogenetic) approach is demonstrated, the clinicians will have at their disposal minimally invasive, longitudinal and follow-up biomarkers, allowing to prevent the emergence of resistance to osimertinib to maintain its effectiveness as longer as possible. It should allow to individualize the dosages for each patient, taking into account their pharmacokinetic profile and the molecular profile of the tumor. This personalized medicine in "2-dimensions" would help to delay tumor progression and would preserve a valuable line of treatment with TKI by optimizing its effectiveness.

The impact of the results of this study is important since the aims are to identify preemptive and predictive biomarkers of drug response and to increase mechanistic knowledge regarding risk factor of resistance to osimertinib. Finally, if the hypotheses evaluated in this translational research study are verified, therapeutic drug monitoring of TKI (and ctDNA analysis) would be immediately applicable in clinical practice since the technical tools are already available in the laboratories of most hospitals centers.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Man or woman
* Diagnosis of locally advanced non-small cell bronchial adenocarcinoma (not eligible for locoregional treatment) or metastatic
* Tumor with an activating mutation of EGF-R (deletion of exon 19 or L858R, L861x, or G719x mutation)
* No one opposed to his participation in the research
* Dated and signed consent form
* Patient in good general condition according to WHO (PS: 0 or 1)

Exclusion Criteria:

* Previous treatment of NSCLC with an EGF-R tyrosine kinase inhibitor
* Adult persons subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.
* Treatment with Osimertinib on going
* Co-treatments with a potent enzyme inducing or inhibitor compound within 2 weeks before starting treatment with Osimertinib
* Participation in intervention research on a drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient naïve to any treatment for the metastatic stage, treated with osimertinib as first line treatment (Prior adjuvant or neoadjuvant treatment with chemotherapy, or radiotherapy, are authorized) with a Diagnosis of locally advanced non-small cell bronchial adenocarcinoma, and followed in one of the investigationnal centers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
relationship between plasma exposure to osimertinib and response to treatment assessed by progression-free survival | at 18 months follow-up
  patients who have not progressed during the first 18 months and those who have progressed during the first 18 months.

SECONDARY OUTCOMES:
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Days 15
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 1
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 2
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 3
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 6
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 9
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month12
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month 15
  ctDNA blood concentration and osimertinib plasma concentration
Longitudinal correlation between the plasma concentration of osimertinib and the concentration of ctDNA (liquid biopsy) | Month18
  ctDNA blood concentration and osimertinib plasma concentration
Correlation between the trough plasma concentration of osimertinib and the time to onset of acquired molecular resistance mutations to osimertinib (identified on ctDNA) | Days 15
  Trough osimertinib plasma concentration and emergence of resistance mutation not present at baseline and / or re-appearance of the of EGF-R baseline mutation on ctDNA
Correlation between the trough plasma concentration of osimertinib and the time to onset of acquired molecular resistance mutations to osimertinib (identified on ctDNA) | At desease progression
  Trough osimertinib plasma concentration and emergence of resistance mutation not present at baseline and / or re-appearance of the of EGF-R baseline mutation on ctDNA
Correlation between the trough plasma concentration of osimertinib and the acquired clinical resistance | Days 15
  Acquired "clinical" resistance (expressed in months) defined as tumor progression (according to RECIST criteria) diagnosed after an initial response period in a patient treated without interruption of osimertinib
Correlation between the trough plasma concentration of osimertinib and the acquired clinical resistance | At desease progression
  Acquired "clinical" resistance (expressed in months) defined as tumor progression (according to RECIST criteria) diagnosed after an initial response period in a patient treated without interruption of osimertinib
Correlation between the concentration of ctDNA and acquired clinical resistance | Days 15
  Acquired "clinical" resistance (expressed in months) and evolution of the blood ctDNA concentration
Correlation between the concentration of ctDNA and acquired clinical resistance | At desease progression
  Acquired "clinical" resistance (expressed in months) and evolution of the blood ctDNA concentration
Study the concentration-toxicity correlation of osimertinib | untill Month 18
  Type and number of grade II to IV adverse events observed under treatment with osimertinib (according to CTCAE V5.0)
Influence of genetic polymorphisms on the plasma concentration of osimertinib (CYP3A4 and ABCB1) | Days 0
  Concentrations of osimertinib in the groups of patients carrying an allelic variant modifying the activity of CYP3A4/5 and / or ABCB1 versus concentrations in the group of patients of wild-type genotype
the inter-individual variability of osimertinib plasma concentration | Days 15
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 1
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 2
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 3
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 6
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 9
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 12
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 15
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the inter-individual variability of osimertinib plasma concentration | Month 18
  Coefficient of variation of trough plasma concentrations of osimertinib between subjects
the intra-individual variability of osimertinib plasma concentration | Days 15
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 1
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 2
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 3
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 6
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 9
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 12
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 15
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period
the intra-individual variability of osimertinib plasma concentration | Month 18
  Coefficient of variation of trough plasma concentrations of osimertinib for the same subject during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Camille TRON, MD, Principal Investigator — Rennes University Hospital
Locations (4):
- France (4):
  - CH Bretagne Sud (Site du Scorff), Lorient
  - Chu de Rennes (Service Pneumologie), Rennes
  - CH Saint Malo (Service de Pneumologie), St-Malo
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Undecided